CLINICAL TRIAL: NCT05934669
Title: Randomized Controlled Trial of Intranasal (IN) Midazolam vs IN Dexmedetomidine vs IN Ketamine Evaluating Length of Stay After Medication Administration and Anxiolysis During Minimal Procedures in Pediatric Population in Pediatric Emergency Department
Brief Title: IN Midazolam vs IN Dexmedetomidine vs IN Ketamine During Minimal Procedures in Pediatric ED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15872
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Laceration of Skin; Anxiety; Discharge Time
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: After patient enrollment, a nurse will assign a chronological number from 1 to 90. The pharmacist will randomly divide all 90 subjects into 3 even groups to receive either medication A, B, or C. The pharmacist will dispense the medication in a 1ml syringe to the chronological number provided in the order. The nurse will fill out a mYPAS scale to assess the patient's anxiety level and then administer the medication. After 30 minutes, the physician will determine subject readiness and perform laceration repair. The patient's vitals will be monitored every 5 minutes. At the end of the procedure, both the physician and the parent will answer a question using a Likert scale and the nurse will fill out another mYPAS scale. After the procedure, the patient will be monitored in the ED for any adverse effects and will be discharged home once the patient meets established discharge criteria. The nurse will document the time the patient is discharged.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double blind randomized study. Except for the pharmacist, all treating ED physicians, nurses, patients, patients' caregivers/guardians, ancillary staff, and data analysts will be blinded to the medication administered to the patient. The medication will be dispensed in a 1ml syringe and the barrel of the syringe will be covered by the pharmacist. All the syringes sent from the pharmacy will appear the same, regardless of the volume of the medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intranasal Midazolam (Experimental): Dose/Concentration: 5mg/ml of 0.4mg/kg Midazolam (max dose 10mg). Adverse side effects include respiratory depression and hypotension. Intranasal Midazolam is standard of care for minimal procedures in pediatric ED.
  Interventions: Drug: Intranasal Midazolam
- Intranasal Dexmedetomidine (Experimental): Dose/Concentration: 100mcg/ml of 2mcg/kg Dexmedetomidine (max dose 100mcg). Adverse side effects include Hypotension and Bradycardia at high dosages. IV Dexmedetomidine is FDA approved and widely used in sedation. IN form isn't FDA approved; however, it has been approved to conduct research studies that have showed its efficacy in pre-operative settings, imaging-CT or MRI, dental procedures, and much more. Specifically, in a pediatric ED setting, Neville et al conducted a study comparing intranasal Dexmedetomidine and intranasal Midazolam prior to laceration repair in a pediatric emergency department and showed safe administration of Dexmedetomidine.
  Interventions: Drug: Intranasal Dexmedetomidine
- Intranasal Ketamine (Experimental): Dose/Concentration: 100mg/ml of 3mg/kg Ketamine (max dose 100mg). Adverse side effect include Laryngospasm. IV Ketamine is FDA approved and widely used in procedural sedation in pediatric EDs. IN form isn't FDA approved in pediatric population; however, it has also been approved to conduct research studies especially in combination with other medications. Gutherie et al conducted a study demonstrating intranasal Ketamine providing safe and successful anxiolysis in pediatric patients in an ED setting.
  Interventions: Drug: Intranasal Ketamine

INTERVENTIONS:
Drug: Intranasal Midazolam — Using a computer-generated randomization schedule by the research pharmacist, all 90 subjects will be divided into 3 even groups to receive either medication A (intranasal Midazolam), B (intranasal Dexmedetomidine), or C (intranasal Ketamine). Based on the randomization schedule, the pharmacist will dispense medication A, B, or C to the chronological number provided in the order. The total amount of the medication will be based on the patient's charted weight. Small volumes of less than 1ml per nostril are preferred for reliable absorption; therefore, the medication will be dispensed in a 1ml syringe and the barrel of the syringe will be covered by the pharmacist. All the syringes sent from the pharmacy will appear the same, regardless of the volume of the medication.
  Other Names: Intranasal Versed
  Arms: Intranasal Midazolam
Drug: Intranasal Dexmedetomidine — See above
  Other Names: Intranasal Precedex
  Arms: Intranasal Dexmedetomidine
Drug: Intranasal Ketamine — See above
  Arms: Intranasal Ketamine

SUMMARY:
Pain in young children has been universally under-recognized due to their inability to describe or localize pain. Improvements in pharmacological interventions are necessary to optimize patient and family experience and allow for successful and efficient procedure completion. This is the first study that will compare three intranasal medications (Intranasal Midazolam, Dexmedetomidine, and Ketamine) to evaluate the length of stay after medication administration along with patient and provider satisfaction. The objective of this study is to demonstrate superior intranasal anxiolysis for pediatric laceration repairs with the shortest emergency department stay and highest patient and provider satisfaction. Based on previous studies and medication pharmacokinetics, we hypothesize that Intranasal Ketamine will have the shortest Emergency Department (ED) stay followed by Midazolam and then Dexmedetomidine with the longest stay; however, Dexmedetomidine will have the highest patient and provider satisfaction followed by Ketamine and then Midazolam.

DETAILED DESCRIPTION:
Children commonly present to ED with injuries requiring procedures that can be painful or require a child to be absolutely still. Pain in young children has been universally under-recognized due to their inability to describe or localize pain. Multiple surveys of parents and families have showed that ED satisfaction is highly dependent on the degree of pain a patient experiences and the efforts made to alleviate the pain. Therefore, improvements in pharmacological interventions are necessary to optimize patient and family experience and allow for successful and efficient procedure completion.

Intranasal Midazolam is widely used for minimal procedural anxiolysis in pediatric population. Intranasal medication delivery has the highest parent and provider satisfaction with the advantage of avoiding painful needle stick and faster absorption compared to oral or intramuscular medication. Midazolam is a gamma-aminobutyric acid (GABA) receptor agonist that can provide anxiolysis and amnesia but no analgesia. Intranasal Midazolam has a rapid onset of 5-10 minutes with peak at 30 minutes. There have been limited studies evaluating the length of stay or time to discharge after medication administration with an average length of stay of about 30 minutes. It has been shown to be safe and effective in children for minor procedures; however, intranasal Midazolam is notoriously noxious and irritating to nasal mucosa and requires larger volumes for intranasal dosing. Main side effects include respiratory depression and hypotension. It is also known to cause paradoxical reaction with hyperactivity, agitation, and restlessness especially in developmentally delayed or children with Autism or behavioral concerns. Therefore, several new studies have evaluated other newer intranasal medications for minor procedures including intranasal Dexmedetomidine and intranasal Ketamine.

Dexmedetomidine is an alpha 2 agonist that mirrors sleep in children and can provide anxiolysis and minimal analgesia. Intranasal dosages that have provided adequate minimal sedation is 2-4mcg/kg (max dosage 100-200mcg) with wide range of onset 10-45 mins with average 30 minutes and peak at 90 minutes. Unlike Midazolam, it preserves airway reflexes without clinically significant hemodynamic instability in children. Studies have also shown that it is well tolerated by children and preferred in children with Autism and behavioral concerns.

Ketamine is an N-methyl-D-aspartate (NMDA) antagonist that provides both anxiolysis and analgesia. It is widely used in ED settings for intravenous procedural sedation; however, intranasal route provides non-invasive method of medication administration. Gutherie et al conducted a study demonstrating intranasal Ketamine providing safe and successful anxiolysis and analgesia in pediatric patients in an ED setting. Intranasal dosage of 3-5mg/kg (max dosage 100-200mg) provides optimal onset of action within 10 minutes with peak at 15-20 minutes and duration of 45-60 minutes. It has few significant side effects including the rare laryngospasm and recovery agitation, however, it preserves airway reflexes and favorable in hemodynamic instability.

Previous Studies:

Limited studies have demonstrated anxiolysis with patient and provider satisfaction or time to discharge after medication administration comparing intranasal Midazolam to intranasal Dexmedetomidine or intranasal Ketamine in a pediatric emergency medicine setting. Neville et al conducted a study comparing intranasal Dexmedetomidine and intranasal Midazolam prior to laceration repair in a pediatric emergency department and concluded that patients who received Dexmedetomidine had less anxiety at the time of positioning for the procedure. Several other studies have demonstrated similar outcomes with better patient and provider satisfaction in pre-operative settings, imaging, and dental settings. Surendar et al is the only study that compared all three intranasal medications. The study included uncooperative pediatric patients in a dental setting. Although overall differences were not statistically significant, the onset of sedation was rapid among Intranasal Ketamine and Midazolam groups but overall success was highest in Dexmedetomidine group.

Objective/Aims/Hypothesis:

This is the first study that will compare all three intranasal medications to evaluate the length of stay after medication administration along with patient and provider satisfaction. The objective of this study is to demonstrate superior intranasal anxiolysis for pediatric laceration repairs with the shortest emergency department stay and highest patient and provider satisfaction. The primary outcome will measure the time to discharge after medication administration. Other measurements with include patient's anxiety using previously validated scale Modified Yale Preoperative Anxiety Scale (mYPAS) and physician and parent satisfaction using 5 point Likert scale. Based on previous studies and medication pharmacokinetics, we hypothesize that Ketamine will have the shortest ED stay followed by Midazolam and then Dexmedetomidine with the longest stay; however, Dexmedetomidine will have the highest patient and provider satisfaction followed by Ketamine and then Midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-5 years old
* Presents to the ED for suture repair for lacerations less than or equal to 5cm in length
* Parent(s)/Caregiver(s) speak English

Exclusion Criteria:

* Younger than 12 months of age or older than 5 years old
* Suture repair needed for lacerations are greater than 5cm in length
* Known allergy or adverse effect to Midazolam, Dexmedetomidine, Ketamine, or any other sedatives
* Any abnormal vital signs for age, especially heart rate and blood pressure
* History of Cardiac, respiratory, renal, or liver disease
* Known electrolyte abnormalities
* Any ocular trauma, nasal injury, nasal deformity, significant nasal congestion, abnormalities in the nasal or oral mucosa, facial deformity, or facial injury
* Home medications include beta blockers or any other blood pressure lowering agents Classified American Society of Anesthesiologists III and above
* Known or anticipated difficult airway
* Abnormal neurological exam
* Parent(s)/Caregiver(s) do not speak English

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will measure the time to discharge after intranasal medication administration | Day 1
  The nurse will document the time the medication is administered and the time of discharge once the patient meets American Academy of Pediatrics (AAP) criteria of discharge. AAP discharge criteria includes cardiovascular function and airway potency satisfactory; arousable and protective reflexes are intact; able to talk appropriately for age; able to sit up appropriately for age; and state of hydration is adequate

SECONDARY OUTCOMES:
The secondary outcome will measure patient's anxiety using the previously validated scale mYPAS and physician and parent satisfaction using a 5-point Likert scale | Day 1
  Once the pharmacy dispenses the medication, the nurse will fill out an 18-point scale survey (Modified Yale Preoperative Anxiety Scale [mYAS]) to assess the patient's anxiety level. At the end of the procedure, both the physician and the parent will answer a question using a 5-point Likert scale and the nurse will fill out the same mYAS survey utilized prior to medication administration. The mYAS scale evaluates four domains including activity, vocalizations, emotional expressivity, and state of apparent arousal. The scoring is combined into a total anxiety score between 23.3 and 100 with a patient scoring less than or equal to 30 being categorized as not anxious. The scores on 5-point Likert scale are categorized into very satisfied, satisfied, no difference, unsatisfied, very unsatisfied for 5, 4, 3, 2, and 1, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mckee, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Research records for this study will be maintained for three years following its completion to allow for inspection by government agencies, the sponsor, the University, and other applicable entities.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three years after the completion of the study

REFERENCES:
- [Background] Shaw KN, Bachur RG, editors. Fleisher & Ludwig's Textbook of Pediatric Emergency Medicine. 8th Edition. Philadelphia: Wolters Kluwer, e129, 2021
- [Background] Zempsky WT, Cravero JP; American Academy of Pediatrics Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine. Relief of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 2004 Nov;114(5):1348-56. doi: 10.1542/peds.2004-1752. PMID 15520120
- [Background] Everitt IJ, Barnett P. Comparison of two benzodiazepines used for sedation of children undergoing suturing of a laceration in an emergency department. Pediatr Emerg Care. 2002 Apr;18(2):72-4. doi: 10.1097/00006565-200204000-00002. PMID 11973494
- [Background] Iirola T, Vilo S, Manner T, Aantaa R, Lahtinen M, Scheinin M, Olkkola KT. Bioavailability of dexmedetomidine after intranasal administration. Eur J Clin Pharmacol. 2011 Aug;67(8):825-31. doi: 10.1007/s00228-011-1002-y. Epub 2011 Feb 12. PMID 21318594
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, Yuen MK. Optimal timing for the administration of intranasal dexmedetomidine for premedication in children. Anaesthesia. 2010 Sep;65(9):922-9. doi: 10.1111/j.1365-2044.2010.06453.x. PMID 20645951
- [Background] Carlone G, Trombetta A, Amoroso S, Poropat F, Barbi E, Cozzi G. Intramuscular Dexmedetomidine, a Feasible Option for Children With Autism Spectrum Disorders Needing Urgent Procedural Sedation. Pediatr Emerg Care. 2019 Jun;35(6):e116-e117. doi: 10.1097/PEC.0000000000001776. No abstract available. PMID 31157751
- [Background] Azizkhani R, Heydari F, Ghazavi M, Riahinezhad M, Habibzadeh M, Bigdeli A, Golshani K, Majidinejad S, Mohammadbeigi A. Comparing Sedative Effect of Dexmedetomidine versus Midazolam for Sedation of Children While Undergoing Computerized Tomography Imaging. J Pediatr Neurosci. 2020 Jul-Sep;15(3):245-251. doi: 10.4103/jpn.JPN_107_19. Epub 2020 Nov 6. PMID 33531939
- [Background] Guthrie AM, Baum RA, Carter C, Dugan A, Jones L, Tackett T, Bailey AM. Use of Intranasal Ketamine in Pediatric Patients in the Emergency Department. Pediatr Emerg Care. 2021 Dec 1;37(12):e1001-e1007. doi: 10.1097/PEC.0000000000001863. PMID 31290798
- [Background] Neville DN, Hayes KR, Ivan Y, McDowell ER, Pitetti RD. Double-blind Randomized Controlled Trial of Intranasal Dexmedetomidine Versus Intranasal Midazolam as Anxiolysis Prior to Pediatric Laceration Repair in the Emergency Department. Acad Emerg Med. 2016 Aug;23(8):910-7. doi: 10.1111/acem.12998. PMID 27129606
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Gyanesh P, Haldar R, Srivastava D, Agrawal PM, Tiwari AK, Singh PK. Comparison between intranasal dexmedetomidine and intranasal ketamine as premedication for procedural sedation in children undergoing MRI: a double-blind, randomized, placebo-controlled trial. J Anesth. 2014 Feb;28(1):12-8. doi: 10.1007/s00540-013-1657-x. Epub 2013 Jun 26. PMID 23800984
- [Background] Surendar MN, Pandey RK, Saksena AK, Kumar R, Chandra G. A comparative evaluation of intranasal dexmedetomidine, midazolam and ketamine for their sedative and analgesic properties: a triple blind randomized study. J Clin Pediatr Dent. 2014 Spring;38(3):255-61. doi: 10.17796/jcpd.38.3.l828585807482966. PMID 25095322
- [Background] Cravero JP, Askins N, Sriswasdi P, Tsze DS, Zurakowski D, Sinnott S. Validation of the Pediatric Sedation State Scale. Pediatrics. 2017 May;139(5):e20162897. doi: 10.1542/peds.2016-2897. PMID 28557732
- [Background] Tug A, Hanci A, Turk HS, Aybey F, Isil CT, Sayin P, Oba S. Comparison of Two Different Intranasal Doses of Dexmedetomidine in Children for Magnetic Resonance Imaging Sedation. Paediatr Drugs. 2015 Dec;17(6):479-85. doi: 10.1007/s40272-015-0145-1. PMID 26323489
- [Background] Marra P, Di Stadio A, Colacurcio V, Scarpa A, La Mantia I, Salzano FA, De Luca P. Sedation with Intranasal Dexmedetomidine in the Pediatric Population for Auditory Brainstem Response Testing: Review of the Existing Literature. Healthcare (Basel). 2022 Feb 1;10(2):287. doi: 10.3390/healthcare10020287. PMID 35206901
- [Background] Lewis J, Bailey CR. Intranasal dexmedetomidine for sedation in children; a review. J Perioper Pract. 2020 Jun;30(6):170-175. doi: 10.1177/1750458919854885. Epub 2019 Jun 27. PMID 31246159